CLINICAL TRIAL: NCT06958497
Title: Safety, Efficacy and Quality of Life of Sphinkeeper Implantation for Fecal Incontinence: Results of Mid-term Follow-up. A Multicenter Retrospective Cohort Study
Brief Title: Safety, Efficacy and Quality of Life of Sphinkeeper Implantation for Fecal Incontinence
Status: Completed | Type: Observational
Sponsor: Academy of Applied Medical and Social Sciences, Poland (Other)
Collaborators: University of Campania Luigi Vanvitelli (Other); Vienna University Hospital, Austria (Unknown); University of Barcelona (Other); St Mark's Hospital Foundation (Other); Imperial College London (Other); The Royal London Hospital, UK (Unknown)
Responsible Party: Principal Investigator, Luigi Marano, Professor, Academy of Applied Medical and Social Sciences, Poland
Other Study IDs: 04002025
Record Dates: First submitted 2025-04-21; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Sphinkeeper™ — The procedure was performed under spinal anesthesia, with the patients in lithotomy position. Ten 2-mm perianal skin incisions were made 1-2 cm from the anal margin (i.e., 0.5-1 cm from the intersphinteral sulcus), equidistant one each other, around the entire anal circumference, to allow implantation of 10 prostheses using a specifically designed delivery system (THD Sphinkeeeper Delivery System, THD Sp, Correggio, Italy). The introducer was placed through each skin incision in the intersphincteric space where the prostheses were delivered at a level below the puborectalis muscle. All of the steps were verified by palpation and direct vision using the Eisenhammer anal speculum. Patients were discharged on the same day and recommended to avoid any trauma or sexual practice during the first 48 hours after implantation. A 5-day course of antibiotics was also prescribed.

SUMMARY:
This study evaluated a treatment called Sphinkeeper™ implantation for people suffering from fecal incontinence, a condition where individuals are unable to control their bowel movements. The procedure involves placing small expandable devices into the anal sphincter area to help improve muscle function and prevent leakage.

Researchers from several European hospitals followed 111 patients over three years to assess how safe and effective this treatment is, and how it affects quality of life. Most patients had not improved with other treatments like diet, medications, or pelvic floor therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults diagnosed with clinical fecal incontinence (FI), defined as experiencing at least one incontinence episode per week for a duration exceeding six months.
* Refractory to all standard conservative treatments, including:

  * Pharmacologic therapy
  * Behavioral interventions
  * Pelvic floor rehabilitation
* Endoanal ultrasonography indicating:

  * Intact internal and external anal sphincters, or
  * Internal, external, or combined sphincter defects involving no more than 120 degrees of the anal circumference.

Exclusion Criteria:

* Presence of inflammatory bowel disease with anorectal involvement.
* Diagnosis of anorectal cancer.
* Evidence of perianal sepsis.
* Endoanal ultrasound detection of sphincter defects extending over more than 120 degrees of the internal or external sphincter, or both.
* Prior treatment with sacral neuromodulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: among all the patients with FI assessed for eligibility, were included in this study the subjects over 18 years of age, affected by clinical FI (defined as at least one incontinence episode per week reported for a period of time longer than six months), who were refractory to all standard conservative measures (pharmacologic, behavioral, and pelvic floor rehabilitation) and who showed, at endosonographic evaluation, intact anal sphincters or internal or external or combined internal and external sphincter defects extending for no more of 120 grades of anal circumference.
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-03 (Actual); Study Completion 2025-03 (Actual)

PRIMARY OUTCOMES:
Change in Number of Fecal Incontinence Episodes per Week | 3 years
  The mean change from baseline in the number of fecal incontinence episodes per week at 3-year follow-up.
  Unit of Measure: Episodes per week
Change in Number of Soiling Episodes per Week | 3 years
  The mean change from baseline in the number of soiling episodes per week at 3-year follow-up.
  Unit of Measure: Episodes per week
Change in Time to Postpone Defecation | 3 years
  The mean change from baseline in the maximum time participants are able to postpone defecation at 3-year follow-up.
  Unit of Measure: Minutes
Change in Cleveland Clinic Incontinence Score (CCIS) | 3 years
  The mean change from baseline in the CCIS at 3-year follow-up. Unit of Measure: Points on the CCIS scale (0-20)
Change in Vaizey Incontinence Score | 3 years
  The mean change from baseline in the Vaizey score at 3-year follow-up. Unit of Measure: Points on the Vaizey scale (0-24)

SECONDARY OUTCOMES:
Change in Fecal Incontinence Quality of Life (FIQoL) Score | 3 years
  Evaluation of the impact of the Sphinkeeper procedure on quality of life, assessed by the Fecal Incontinence Quality of Life (FIQoL) Scale.
  The FIQoL Scale consists of 29 items across four domains (Lifestyle, Coping/Behavior, Depression/Self-Perception, Embarrassment).
  Each item is scored from 1 to 4, with higher scores indicating a better quality of life.
  Domain scores and a total score are calculated; higher scores reflect better functioning and reduced impact of fecal incontinence.
  Unit of Measure: Points on the FIQoL Scale (range: 1-4 per item; total scores vary depending on domain aggregation).

IPD SHARING:
Plan to Share IPD: Undecided